CLINICAL TRIAL: NCT00985244
Title: Influence of Macrolide Maintenance Therapy and Bacterial Colonisation on Exacerbation Frequency and Progression of COPD, a Randomized Double-blind Placebo-controlled Trial
Brief Title: Macrolide Maintenance Therapy in Chronic Obstructive Pulmonary Disease
Acronym: COLUMBUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R.S. Djamin (Other)
Collaborators: Erasmus Medical Center (Other); Stichting Solong (Unknown); Amphia Hospital (Other)
Responsible Party: Sponsor-Investigator, R.S. Djamin, MD, Amphia Hospital
Organization: Amphia Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Amphia-ABR29500; 2009-015857-19 (EudraCT Number)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: COPD
Keywords: COPD; COPD exacerbation; macrolide; diseae progression; bacterial colonisation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin (Active Comparator): Subjects in this group will receive 3 times a week 500 mg of the antibiotic azithromycin
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Subjects in this group will receive 3 times a week placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Subjects in this group will receive 3 times a week 500 mg of the antibiotic azithromycin during 1 year.
  Other Names: Zithromax; Azitrocin; Ultreon; Azadose; Sumamed; Azacleus; Nuzaca; Toraseptol; Vinzam; Zentavion
  Arms: Azithromycin
Drug: Placebo — Persons in this group will receive 3 times a week placebo of azithromycin during 1 year.
  Arms: Placebo

SUMMARY:
To assess whether maintenance treatment with macrolide antibiotics in COPD patients with three or more exacerbations in the preceding year of inclusion can decrease the exacerbation rate in the year of treatment.

DETAILED DESCRIPTION:
COPD is characterized by progressive development of airflow limitation that is poorly reversible. Because of a poor understanding of COPD pathogenesis, treatment is mostly symptomatic and new therapeutic strategies are limited. There is a direct relationship between the severity of the disease and the intensity of the inflammatory response.One of the hypothesis for persistent airway inflammation is that the presence of recurrent infections is responsible for this condition.

Macrolide antibiotics have a bacteriostatic as well as anti-inflammatory properties. This clinical trial will investigate whether maintenance treatment with macrolide antibiotics during 1 year in people with 3 or more exacerbations in the preceding year of inclusion can decrease the exacerbation rate in that same year of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD according to GOLD criteria (FEV1/FVC<70%), classification into GOLD I (FEV1 70-100% predicted), GOLD II (FEV1 50-70% predicted), GOLD III (FEV1 30- 50% predicted) or GOLD IV (FEV1 ≤ 30% predicted)
* Age ≥ 18 years
* Three or more exacerbations of COPD in one year for which a course of prednisone and/or antibiotic therapy was started
* Clinically stable during 1 month. Patients have to be free of COPD exacerbation or respiratory tract infection within a month prior to involvement in the study and they should not have received a high dose of systemic glucocorticoids or antibiotics in this period
* Informed consent

Exclusion Criteria:

* Use of antibiotics or high dose of systemic steroids within a month prior to involvement in the study.
* Addition of inhalation steroids to the patient's therapy regimen, shortly before entering the study.
* Pregnant or lactating women.
* Allergy to macrolides.
* Liver disease (alanine transaminase and/or aspartate transaminase levels 2 or more times the upper limit of normal).
* Asthma, defined as episodic symptoms of airflow obstruction which is reversible with bronchodilators, assessed with lung function testing.
* Presence of a malignancy which is clinically active.
* Bronchiectasis.
* Malignancy of any kind for which the subject is under treatment or is being monitored as part of follow up after treatment.
* Heart failure.
* Use of drugs which can adversely interact with macrolides and for which therapeutic monitoring cannot be undertaken.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Reduction in number of exacerbations | 1 year

SECONDARY OUTCOMES:
Lung function parameters (FEV1 (L), FVC (L), FRC (L), RV (L), TLC(L), IC (L), 6 minute walking distance) | Day 1. Also 3, 6, 9 and 12 months.
Disease specific health related quality of life measured by St. George's Respiratory Questionnaire (SGRQ) | Day 1. Also 3, 6, 9 and 12 months. In case of an exacerbation.
Indication of anxiety and depression by Hospital Anxiety Depression Scale (HADS) | Day 1. Also 3, 6, 9 and 12 months.
Microbiology of sputum (culture and PCR). | Day 1. Also 3, 6, 9 and 12 months. In case of an exacerbation of COPD.
Measurement of inflammatory markers in sputum and serum. | Day 1. Also 3, 6, 9 and 12 months. In case of an exacerbation of COPD.
Adverse events of treatment. | Day 1. Also 3, 6, 9 and 12 months. Whenever adverse events occur.
Length of hospital stay. | Whenever admission to hospital is required for an exacerbation of COPD.
Time till next exacerbation. | Whenever an exacerbation of COPD occurs.
Assess type D personality by DS-14 questionnaire. | Day 1 and month 12.
Generic health status measured by 12-Item Short Form Health Survey (SF-12). | Day 1, month 3, 6, 9 and 12. In case of an exacerbation.
Decrease in percentage of clinical versus outdoor department exacerbations. | Month 12.
Effect of maintenance macrolides on intestinal bacterial restistancy patterns | Day 1, month 6 and month 12
Serology and PCR for atypical microorganisms in serum | day 1. In case of an exacerbation.
Intestinal bacterial resistance patterns | Day 1, month 6 and month 12
  Rectal swabs will be tested for bacterial resistance patterns and change in rectal flora as a result of maintenance azithromycin.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Aerts, MD, PhD, Study Director — Amphia ziekenhuis; Menno van der Eerdem, MD, PhD, Study Director — Erasmus Medical Center
Locations (1):
- Amphia Ziekenhuis, Breda, North Brabant, Netherlands

REFERENCES:
- [Derived] Djamin RS, Talman S, Schrauwen EJA, von Wintersdorff CJH, Wolffs PF, Savelkoul PHM, Uzun S, Kerstens R, van der Eerden MM, Kluytmans JAJW. Prevalence and abundance of selected genes conferring macrolide resistance genes in COPD patients during maintenance treatment with azithromycin. Antimicrob Resist Infect Control. 2020 Jul 28;9(1):116. doi: 10.1186/s13756-020-00783-w. PMID 32723393
- [Derived] Uzun S, Djamin RS, Kluytmans JA, Mulder PG, van't Veer NE, Ermens AA, Pelle AJ, Hoogsteden HC, Aerts JG, van der Eerden MM. Azithromycin maintenance treatment in patients with frequent exacerbations of chronic obstructive pulmonary disease (COLUMBUS): a randomised, double-blind, placebo-controlled trial. Lancet Respir Med. 2014 May;2(5):361-8. doi: 10.1016/S2213-2600(14)70019-0. Epub 2014 Apr 15. PMID 24746000
- [Derived] Uzun S, Djamin RS, Kluytmans J, Van't Veer NE, Ermens AA, Pelle AJ, Mulder P, van der Eerden MM, Aerts J. Influence of macrolide maintenance therapy and bacterial colonisation on exacerbation frequency and progression of COPD (COLUMBUS): study protocol for a randomised controlled trial. Trials. 2012 Jun 9;13:82. doi: 10.1186/1745-6215-13-82. PMID 22682323